CLINICAL TRIAL: NCT04819828
Title: Tamsulosin as Adjunctive Therapy After Extracorporeal Shock Wave Lithotripsy for Renal Stones
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Regional de Alta Especialidad del Bajio (Other)
Responsible Party: Principal Investigator, Rafael Maldonado-Valadez, MD, MSc, Hospital Regional de Alta Especialidad del Bajio
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CI-HRAEB-2008-009
Record Dates: First submitted 2021-03-25; First posted 2021-03-29 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Renal Stone
Keywords: Extracorporeal shock wave lithotripsy; Tamsulosin; Urolithiasis
MeSH Terms: conditions — Nephrolithiasis; Urolithiasis | interventions — Lithotripsy; Diclofenac; Tamsulosin

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tamsulosin (Experimental): At the end of the ESWL session, the patients received standard treatment for analgesia consisting of oral diclofenac (75 mg/12 h) as needed plus oral tamsulosin (0.4 mg/day) for eight weeks.
  Interventions: Procedure: Extracorporeal shock wave lithotripsy; Drug: Diclofenac; Drug: Tamsulosin
- Control (Active Comparator): At the end of the ESWL session, the patients received standard treatment for analgesia consisting of oral diclofenac (75 mg/12 h) as needed
  Interventions: Procedure: Extracorporeal shock wave lithotripsy; Drug: Diclofenac

INTERVENTIONS:
Procedure: Extracorporeal shock wave lithotripsy — A single session of extracorporeal shock wave lithotripsy: the session will be finished upon reaching a maximum of 4,000 shocks or if a complete fragmentation of the kidney stone is observed.
Drug: Diclofenac — Standard treatment for analgesia: oral diclofenac (75 mg/12 h) as needed.
Drug: Tamsulosin — Oral tamsulosin (0.4 mg/day) for eight weeks.
  Arms: Tamsulosin

SUMMARY:
Urolithiasis is a common health problem worldwide affecting approximately 10% of the population at some stage in their lives. The aim of this study is to evaluate the efficacy of adjuvant treatment with tamsulosin for improving the stone-free rate after a single session of extracorporeal shock wave lithotripsy (ESWL) in the treatment of radiopaque kidney stones.

DETAILED DESCRIPTION:
Urolithiasis is a common health problem worldwide affecting ∼10% of the population at some stage in their lives. It affects approximately 5% of women and 12% of men in the United States, and it has been suggested that the incidence is increasing. Because of its efficacy and low morbidity, extracorporeal shock wave lithotripsy (ESWL) is an effective treatment for kidney stones smaller than 20 mm in diameter. The objective of this therapy is to achieve an adequate fragmentation of the calculus that allows a spontaneous expulsion of the fragments, and finally, a stone-free state, which is not always possible.

The presence of adrenergic receptors in the ureter has suggested the involvement of the sympathetic nervous system in its peristaltic activity. It has also been shown that alpha 1 adrenergic antagonist medications such as tamsulosin are capable of inhibiting the basal tone and the ureteral peristalsis, causing dilation and facilitating the migration of stones. Some authors have reported the efficacy of this type of medication for spontaneous calculus expulsion, but there is no conclusive evidence of the adjuvant effectiveness of tamsulosin after ESWL for stone clearance and even less among a Mexican population.

This is a single center, randomized, non-placebo-controlled study with a sample of adults (men and women ≥18 years old) with a single radiopaque kidney stone (5-20 mm) in diameter. Post-ESWL session, the patients will be randomly divided into two groups (the control group and the tamsulosin group). After discharge, all patients will be instructed to drink a minimum of 2 L water daily. The control group will receive standard treatment for analgesia consisting of oral diclofenac (75 mg/12 h) as needed. The tamsulosin group will receive standard treatment for analgesia plus oral tamsulosin (0.4 mg/day) for eight weeks.

Patients will attend follow-up visits every two weeks during the first month of treatment and a final visit at the end of the second month. During each visit, vital signs will be taken, a physical examination will be conducted, and possible adverse effects will be monitored; additionally, a plain X-ray of the kidney, ureter, and bladder (KUB) will be taken at two and four weeks for evaluating possible complications associated with residual fragments, as well as an abdominal CT scan at eight weeks after the ESWL in order to determine stone-free status.

Data will be analyzed using R Statistical Software. Descriptive statistics will be determined for the patients' clinical characteristics, grouped by the treatment assigned (control group and tamsulosin group) and will be compared using the Mann-Whitney U test or the chi-square test depending on the variable type. The strength of the association between the ESWL treatment with adjuvant tamsulosin and the stone-free rate will be evaluated by calculating the relative risk (RR) and the number needed to treat (NNT). In all cases, an alpha=0.05 was considered significant.

ELIGIBILITY:
Inclusion Criteria:

* A single radiopaque kidney stone (5-20 mm) in diameter visible on CT scan of the abdomen.

Exclusion Criteria:

* A lower calyx stone.
* A history of spontaneous stone passage.
* A previous failed ESWL.
* Treatment with alpha adrenergic antagonists, calcium channel inhibitors or steroids.
* Severe obesity (BMI≥40).
* Pregnancy.
* Serum creatinine ≥2 mg/dl.
* Renal artery aneurysm and/or abdominal aorta aneurysm.
* The presence of a ureteral stent.
* Anatomical abnormalities or previous surgery on the upper urinary tract.
* Bone deformities.
* Presence of a urinary tract infection.
* Coagulation disorders.
* Poorly controlled hypertension.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2010-01-01 (Actual); Primary Completion 2016-08-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Stone-free rate | 8 weeks
  Percentage of patients with the absence of residual stones (≥ 5 mm in diameter), with the presence of asymptomatic nonsignificant residual stone fragments (≤4 mm in diameter) determined via abdominal computed tomography scan, and with the absence of additional procedures to resolve an event of acute symptomatic urinary obstruction.

SECONDARY OUTCOMES:
Complications rate associated with residual stone fragments | 2, 4, and 8 weeks
  Percentage of patients with the presence of complications associated with residual stone fragments.

CONTACTS AND LOCATIONS:
Overall Officials: Rafael E Maldonado-Valadez, MD, MSc, Principal Investigator — Hospital Regional de Alta Especialidad del Bajio; Edel R Rodea-Montero, MPH, Study Chair — Hospital Regional de Alta Especialidad del Bajio; Jose A Alvarez-Canales, MD, Phd, Study Chair — Hospital Regional de Alta Especialidad del Bajio; Angel D Valdez-Vargas, MD, Study Chair — Hospital Regional de Alta Especialidad del Bajio

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Maldonado-Valadez RE, Valdez-Vargas AD, Alvarez JA, Rodea-Montero ER. Efficacy of Adjuvant Tamsulosin for Improving the Stone-Free Rate after Extracorporeal Shock Wave Lithotripsy in Renal Stones: A Randomized Controlled Trial. Int J Clin Pract. 2022 Jan 31;2022:3757588. doi: 10.1155/2022/3757588. eCollection 2022. PMID 35685573